CLINICAL TRIAL: NCT05051254
Title: Respiratory Muscles and Work of Breathing in Children
Acronym: WOB&MR_Ped
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210261; ID-RCB 2020-A03393-36 (Other: ID RCB Number)
Record Dates: First submitted 2021-06-14; First posted 2021-09-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Neuromuscular Diseases; Congenital Diaphragmatic Hernia; Lung Diseases; Cardiac Diseases; Scoliosis; Diaphragmatic Impairment; Respiratory Muscle Impairment
Keywords: Respiratory muscle testing; Respiratory muscle strength; Work of breathing; Esogastric pressures; Diaphragmatic dysfunction; Diaphragmatic paralysis
MeSH Terms: conditions — Neuromuscular Diseases; Hernias, Diaphragmatic, Congenital; Lung Diseases; Heart Diseases; Scoliosis; Respiratory Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Respiratory muscle impairment (Experimental): Minor patients with primary or secondary impairment of respiratory muscles and followed at Necker Hospital
  Interventions: Other: Esogastric pressure measurement

INTERVENTIONS:
Other: Esogastric pressure measurement — Measurement of work of breathing and respiratory muscles strength using an esogastric catheter.
  One measurement or before and after (6 months and 1 year) the initiation of a pharmacological treatment in order to assess the effect of the treatment on respiratory muscle function.

SUMMARY:
Respiratory muscle testing allows a quantitative assessment of inspiratory and expiratory muscles in children of any age with primary or secondary respiratory muscle impairment, in order to better understand the pathophysiology of respiratory impairment and guide therapeutic management. The use of an invasive technique (esogastric probe) makes it possible to specifically explore the diaphragm, the accessory inspiratory muscles and the expiratory muscles in order to detect dysfunction or paralysis of these muscles, and to estimate the work of breathing in order to better guide the respiratory management.

The primary objective of the study is to evaluate the respiratory effort in children with primary or secondary impairment of the respiratory muscles during spontaneous breathing or during mechanical ventilation.

DETAILED DESCRIPTION:
Respiratory muscle testing allows a quantitative assessment of inspiratory and expiratory muscles in children of any age with primary or secondary respiratory muscle impairment, in order to better understand the pathophysiology of respiratory impairment and guide therapeutic management. The use of an invasive technique (esogastric probe) makes it possible to specifically explore the diaphragm, the accessory inspiratory muscles and the expiratory muscles in order to detect dysfunction or paralysis of these muscles, and to estimate the work of breathing in order to better guide the respiratory management.

Respiratory muscle testing by means of esogastric measurements may allow assessing the effect of pharmacological treatment by comparing respiratory muscle strength before and after a few months with treatment. Moreover, esogastric measurements can be used to better adapt mechanical ventilation or to determine the possibility of weaning from the respiratory support.

The primary objective of the study is to evaluate the respiratory effort in children with primary or secondary impairment of the respiratory muscles during spontaneous breathing or during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than 18 years old with primary or secondary impairment of respiratory muscles and followed at Necker Hospital
* Patients under spontaneous breathing or noninvasive or invasive mechanical ventilation
* Written informed consent

Exclusion Criteria:

* No social insurance
* Significant psychomotor retardation
* Absence of cooperation
* Significant agitation
* Hemodynamic instability
* Acute condition or temporary drug treatments that may interfere with the results of the respiratory muscle explorations

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 550 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Esophageal pressure-time product (PTPoes) | Day 0
  The integral of the esophageal pressure signal over inspiratory time
Diaphragmatic pressure-time product (PTPdi) | Day 0
  The integral of the transdiaphragmatic pressure signal over inspiratory time
Work of breathing (WOB) | Day 0
  Total work of breathing (WOBt) is calculated (in Joules/L) as the area under the pressure-volume curve, using the Campbell diagram. Elastic (WOBe) and resistive (WOBr) are estimated as the 2/3 and 1/3 of WOBt value, respectively.

SECONDARY OUTCOMES:
Vital capacity | Day 0
  Vital capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation, using spirometry
Maximal respiratory static pressures | Day 0
  Maximal static inspiratory and expiratory airway pressures
Maximal sniff pressure | Day 0
  Airway pressure during a sniff test
Maximal whistle pressure | Day 0
  Airway pressure during a whistle test
Peak expiratory flow | Day 0
  Maximal flow during expiratory maneuver
Peak cough flow | Day 0
  Maximal flow during cough
Esophageal pressure during sniff | Day 0
  Esophageal pressure measurement during a sniff test
Gastric pressure during sniff | Day 0
  Gastric pressure measurement during a sniff test
Transdiaphragmatic pressure during sniff | Day 0
  Transdiaphragmatic pressure measurement during a sniff test
Crying transdiaphragmatic pressure | Day 0
  Transdiaphragmatic pressure measurement during crying in young children
Gastric pressure during cough | Day 0
  Gastric pressure measurement during a maximal cough maneuver
Twitch transdiaphragmatic pressure | Day 0
  Transdiaphragmatic pressure measurement during cervical magnetic stimulation
Inspiratory muscles tension-time index | Day 0
  Measurement of the tension-time index of the inspiratory muscles
Diaphragmatic tension-time index | Day 0
  Measurement of the tension-time index of the diaphragm
Correlation between the pressure-time product, the work of breathing and the respiratory muscle strength with the disease severity | Day 0
  The pressure-time product of the respiratory muscles, the work of breathing and the respiratory muscle strength will be correlated with disease severity
Correlation between the pressure-time product, the work of breathing and the respiratory muscle strength with polysomnography and gas exchange results | Day 0
  The pressure-time product of the respiratory muscles, the work of breathing and the respiratory muscle strength will be correlated with the polysomnography and gas exchange results
Esophageal pressure-time products in patients with any treatment and in patients with no treatment | Day 0
  The esophageal pressure-time product will be compared between patients with any treatment and patients receiving no treatment
The total work of breathing in patients with any treatment and in patients with no treatment | Day 0
  The total work of breathing (WOBt), which is calculated (in Joules/L) as the area under the pressure-volume curve using the Campbell diagram, be compared between patients with any treatment and patients receiving no traeatment, using the Student t test
Measurement of esophageal pressure during a sniff in patients with any treatment and patients with no treatment | Day 0
  The esophageal pressure during a sniff will be compared between patients with any treatment and patients receiving no treatment
Measurement of the esophageal pressure-time product before and after pharmacological treatment | 6 months and 1 year after treatment initiation
  The esophageal pressure-time product will be compared before treatment, and 6 months and 1 year after pharmacological treatment initiation
The total work of breathing before and after pharmacological treatment | 6 months and 1 year after treatment initiation
  The total work of breathing (WOBt), which is calculated (in Joules/L) as the area under the pressure-volume curve using the Campbell diagram, will be compared before treatment, and 6 months and 1 year after pharmacological treatment initiation, using the ANOVA on repeated measures
Measurement of the esophageal pressure during a sniff before and after pharmacological treatment | 6 months and 1 year after treatment initiation
  The esophageal pressure during a sniff will be compared before treatment, and 6 months and 1 year after pharmacological treatment initiation
Measurement of transdiaphragmatic pressure during a sniff before and after pharmacological treatment | 6 months and 1 year after treatment initiation
  The transdiaphragmatic pressure measurement during a sniff will be compared before treatment, and 6 months and 1 year after pharmacological treatment initiation
Adaptation of the respiratory support according to the esophageal pressure-time product values | Day 0
  The esophageal pressure-time product will be measured to guide the respiratory support adaptation
Adaptation of the respiratory support according to the total work of breathing values | Day 0
  The total work of breathing (WOBt), which is calculated (in Joules/L) as the area under the pressure-volume curve using the Campbell diagram, will be measured to guide the respiratory support adaptation
Measurement of the esophageal pressure-time product in patients with weaning success and in patients with weaning failure | Day 0
  The esophageal pressure-time product will be compared between patients with weaning success and weaning failure
Measurement of the total work of breathing in patients with weaning success and in patients with weaning failure | Day 0
  The total work of breathing (WOBt), which is calculated (in Joules/L) as the area under the pressure-volume curve using the Campbell diagram, will be compared between patients with weaning success and weaning failure, using the Student t test
Measurement of the esophageal pressure during a sniff in patients with weaning success and in patients with weaning failure | Day 0
  The esophageal pressure during a sniff will be compared between patients with weaning success and weaning failure
Correlation between the pressure-time product, the work of breathing and the respiratory muscle strength with the gas exchange during weaning trial | Day 0
  The pressure-time product, the work of breathing and the respiratory muscle strength will be correlated with the gas exchange during a weaning trial

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte FAUROUX, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Sonia KHIRANI, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No